CLINICAL TRIAL: NCT06147713
Title: Vibrotactile Foot Device for Freezing of Gait in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vibrotactile Foot Device
Record Dates: First submitted 2023-11-14; First posted 2023-11-28 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Freezing of Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The subjects will be examined during the drug-off period with the vibrotactile foot device off and on at different patterns. The tests will be carried out during the onsite clinical visits on the day of initial enrollment and two weeks after home wearing.
  Interventions: Device: Vibrotactile foot device (Smart shoe)

INTERVENTIONS:
Device: Vibrotactile foot device (Smart shoe) — A foot device deliver vibrotactile stimulation triggered by a foot pressure sensor.

SUMMARY:
Freezing of gait (FOG) is a common, disabling symptom of later stage Parkinson's disease (PD), and can induce significant morbidity and mortality by increasing risk of falls as the disease progresses. Despite optimum medical management and deep brain stimulation therapy, many patients with PD are incapacitated by FOG and gait disorders. Non-invasive vibrotactile stimulation has been reported to potentially improve FOG of patients with PD. However, results of studies were variable, and there is a lack of convenient vibrotactile devices ready for daily use with reliable clinical trial data. In the proposed study, the investigator will test the effect of a newly developed vibrotactile foot device (Smart shoe) on participants diagnosed with PD and FOG. EEG and fMRI are obtained in order to investigate the underlying neurological mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years
* Diagnosed with Parkinson's Disease according to MDS Clinical Diagnostic Criteria
* Stable drug therapy without any change in the past one month
* Subjective presence of FOG more than once per day
* Objective presence of FOG by provoking tasks, e.g., gait initiation, rapid full turn, et al.
* Able to walk unaided at least 20 meters
* Provide written informed consent

Exclusion Criteria:

* Stroke and other diseases interfering ambulation
* Severe foot sensory impairments disabling the individual to perceive vibratory stimulation
* History of deep brain stimulation surgery

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
New Freezing of Gait Questionnaire (NFOGQ) | 2 weeks
  Changes in the New Freezing of Gait Questionnaire (NFOGQ) score
Freezing severity | 2 weeks
  Changes in the quantified freezing severity during walking task, videotape reviewed by movement disorder specialists

SECONDARY OUTCOMES:
Quantitative Gait parameters | 2 weeks
  Changes in gait parameters such as stride length, et al. during walking tasks
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | 2 weeks
  Changes in the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III score
Berg Balance Scale | 2 weeks
  Changes in the Berg Balance Scale score
Number of falls and near falls | 2 weeks
  Changes in number of falls and near falls during intervention period
39-item Parkinson's Disease Questionnaire (PDQ-39) | 2 weeks
  Changes in the 39-item Parkinson's Disease Questionnaire (PDQ-39) score
Clinical Global Impressions Scale (CGI-I) | 2 weeks
  Changes in the Clinical Global Impressions Scale (CGI-I) score

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, China